CLINICAL TRIAL: NCT06103370
Title: Syringe Service Based Telemedicine and Social Network Driven HIV Prevention Service Implementation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Maryland Department of Health and Mental Hygiene (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00374291; R01DA058387 (NIH)
Record Dates: First submitted 2023-10-23; First posted 2023-10-26 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections; Substance Use Disorders; Addiction; Opioid Use; Drug Use; Intravenous Drug Usage
Keywords: Injection Drug Use; HIV Prevention; Social Networks
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-educator-based network intervention (Experimental): Indexes randomized to the intervention arm will complete a training program that emphasizes effective communication, frequent HIV testing, and awareness of evidence-based HIV prevention and treatment services. An important innovation to the network intervention will be training indexes to use and distribute HIV self-test kits and naloxone to their network members (NMs).
  Interventions: Behavioral: Peer-educator-based network
- Equal-attention control (No Intervention): This group will receive training sessions that will be focused on the opioid overdose epidemic and will not include any training to serve as a peer educator.

INTERVENTIONS:
Behavioral: Peer-educator-based network — The intervention is a social network-based method of dispersing HIV knowledge, HIV self-testing (HIVST) kits, and naloxone in social networks of people who inject drugs (PWID). It targets index participants (peers) to receive training on HIVST, peer education, and linkage to syringe service programs (SSPs) for HIV services.
  Arms: Peer-educator-based network intervention

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a social network intervention to recruit people who inject drugs and their networks for HIV testing and linkage to HIV prevention and treatment services in Maryland. Study aims are to determine the effectiveness of a social network driven intervention to increase:

* HIV testing (primary);
* PrEP knowledge;
* Uptake of HIV services and pre-exposure prophylaxis (PrEP);
* Uptake of medication for opioid use disorder (MOUD) initiation.

Eligible participants who access syringe service programs (SSPs) serving two counties in Maryland and their risk network members (NMs) will be recruited using an established network inventory and coupon recruitment method. When an index successfully recruits NMs, the index-NM cluster will be randomized to either a peer-educator intervention arm or an equal-attention control arm. Index participants randomized to the peer-educator intervention arm will complete a training program adapted with stakeholder input to context that emphasizes effective communication, frequent HIV testing, and awareness of evidence-based HIV prevention and treatment services. An important innovation to the network intervention will be training indexes to use and distribute HIV self-test kits and naloxone to their NMs. Index participants randomized to the equal-attention control arm will receive training sessions focused on the opioid overdose epidemic and will not include any training to serve as a peer educator. All participants (indexes and NMs) will complete study assessments at baseline and at 3 and 9 months. We will compare the peer-educator intervention group and the equal-attention control group on rates of HIV testing, knowledge of PrEP options and resources, and rates of initiation of HIV treatment, PrEP, and MOUD treatment since the previous assessment (past 3 or 6 months).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for index participants:

* Aged 18 or older
* Self-reported injection drug use in the prior month
* Accessed services at the SSP in the prior 3 months
* Willing to undergo training and attend weekly booster group sessions
* Able to recruit at least 1 drug use Network Member (NM) into study
* Willing to talk with peers about PWID topics such as HIV prevention and care
* Not previously enrolled in the study as index or NM
* English-speaking

Inclusion criteria for network member participants:

* Aged 18 or older
* Self-reported injection drug use in the prior month
* Have a valid coupon or able to recall the 3-digit ID number
* Not previously enrolled in the study as index or NM
* English-speaking

Exclusion criteria:

• Individuals lacking the capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of HIV testing for Network Members | 3 months, 9-months
  Proportion of Network Members (both study arms) who report that they conducted HIV testing since the previous study assessment (i.e., in the prior 3 or 6 months).

SECONDARY OUTCOMES:
Proportion of HIV testing for Index and Network Members | 3- and 9-month follow-up
  Proportion of Index and Network Members (both study arms) who report testing since the previous study assessment (i.e., in the prior 3 or 6 months).
Proportion of HIV testing for Index Members | 3- and 9-month follow-up
  Proportion of Index Members (both study arms) who report testing since the previous study assessment (i.e., in the prior 3 or 6 months).
Proportion of HIV negative participants who have used PrEP | 3- and 9-month follow-up
  Proportion of HIV-negative participants who have used PrEP (yes/no) since the previous study assessment (i.e., in the prior 3 or 6 months) among Network Members.
Change in Knowledge of PrEP options | 3- and 9-month follow-up
  Knowledge of PrEP options and resources measured by questionnaire at 3 and 9 months among Network Members.
Proportion of participants using anti-retroviral therapy (ART) | 3- and 9-month follow-up
  Proportion of participants living with HIV who reported they are currently using anti-retroviral therapy (ART), (yes/no) at the 3- or 9-month follow-up among Network Members.
Proportion of participants who have used Medication for opioid use disorder (MOUD) uptake | 3- and 9-month follow-up
  Proportion of participants who report that they have used MOUD (yes/no) since the previous study assessment (i.e., in the prior 3 or 6 months) among Network Members.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwaseun Falade-Nwulia, MBBS, MPH, Principal Investigator — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Frederick County Health Department, Street Safe Program, Frederick, Maryland

IPD SHARING:
Plan to Share IPD: No